CLINICAL TRIAL: NCT02568605
Title: Prebiotic Fibre Supplementation and Gut Microbiota in Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UC-REB14-2464
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: Dietary intervention; Prebiotic fibre; Weight loss; Gut microbiota; Obesity; Liver fat; Hepatic fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Weight Loss; Obesity; Fatty Liver; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prebiotic Fibre (Experimental): The intervention group will receive two 8g packets/day of prebiotic fibre to add to 250 ml of water and consume 30 minutes prior to breakfast and dinner.
  Interventions: Dietary Supplement: Prebiotic fibre; Behavioral: Weight Loss
- Placebo (Placebo Comparator): The control group will receive two 3g packets/day of maltodextrin to add to 250 ml of water and consume 30 minutes prior to breakfast and dinner.
  Interventions: Dietary Supplement: Placebo; Behavioral: Weight Loss
- Weight Loss (Other): All participants will be supported through Registered Dietitian visits to achieve approximately 10% weight loss.
  Interventions: Behavioral: Weight Loss

INTERVENTIONS:
Dietary Supplement: Prebiotic fibre — Oligofructose-enriched inulin (Synergy1)
  Arms: Prebiotic Fibre
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo
Behavioral: Weight Loss — All participants will receive 10 one-on-one sessions with a Registered Dietitian designed to achieve 10% weight loss over 6 months. The sessions will focus on nutrition education and behavior counseling to reduce food intake and improve dietary quality.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a condition where accumulation of fat in the liver leads to metabolic dysfunction. Currently there are no approved treatments for NAFLD. Part of the metabolic dysfunction may arise through changes in the gut microbiota. Prebiotic fibres have beneficial effects on glucose tolerance, body weight, and gut microbiota; therefore they may have potential as part of a dietary strategy for NAFLD treatment.

DETAILED DESCRIPTION:
The main objective of this study is to assess the effect of prebiotic fibre supplementation, in conjunction with diet-induced weight loss, on reduction in liver fat and injury.

Primary Objective - determine the change in hepatic injury (fibrosis and inflammation) and hepatic fat (percent fat) over 6 months in NAFLD patients treated with prebiotic or placebo during weight loss.

Secondary Objectives - determine the changes in appetite, body composition, glycemic and insulinemic responses, quality of life with prebiotic or placebo during weight loss, and examine mechanisms related to prebiotic-induced changes in gut microbiota and lipogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects diagnosed with NAFLD on the basis of abnormal liver enzymes (ALT>1.5x upper limit of normal) and ultrasonography
* Exclusion of other causes of liver disease including viral hepatitis and alcoholic liver disease
* Aspartate aminotransferase and alanine aminotransferase ≤10x upper limit of normal
* Patients with type 2 diabetes treated with diet and exercise alone or metformin

Exclusion Criteria:

* Cirrhosis of the liver (FibroScan >17.5 kilopascal or FibroTest >0.8) or clinical features of cirrhosis.
* Alcohol consumption >20g/day (2 standard drinks) in women or > 30g/d (3 drinks) in men
* Alternate (e.g. TPN) or concomitant etiology for abnormal liver enzymes.
* History of decompensated liver disease including ascites, encephalopathy or variceal bleeding
* Concomitant use of any weight loss medication, previous bariatric or other intestinal surgery
* Presence of active infection, pregnancy or lactation
* Regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment
* Antibiotic use within 3 months prior to enrollment
* Weight loss >3 kg within preceding 3 months to enrollment
* Uncontrolled cardiovascular or respiratory disease, active malignancy, or chronic infections
* Use of agents such as vitamin E, omega-3 fatty acids or medications with evidence for effects on NAFLD (pioglitazone, Glucagon-like peptide-1 analogues, dipeptidyl peptidase IV inhibitors, ursodeoxycholic acid)
* Patients with type 2 diabetes where HbA1c is >9%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Change in Liver Fat | 24 weeks
  Assessed via MRI
Change in Liver Fibrosis | 24 weeks
  Assessed via FibroScan (transient elastography)
Change in Liver Injury | 24 weeks
  Assessed via Fibrotest Score (composite score from serum biochemical markers: alfa2-macroglobulin, apolipoproteinA1, total bilirubin, haptoglobin, gamma glutamyl transpeptidase, alanine aminotransferase)

SECONDARY OUTCOMES:
Change in Glucose Tolerance | 24 weeks
  Assessed via an oral glucose tolerance test
Change in Glycemic Control | 24 weeks
  Assessed via HbA1c
Change in Subjective Appetite | 24 weeks
  Assessed via Subjective appetite ratings on a visual analogue scale
Change in Satiety Hormones | 24 weeks
  Assessed in serum as pg/ml (Ghrelin, Glucagon-like peptide-1, Glucose-dependent insulinotropic polypeptide, leptin and Peptide tyrosine tyrosine)
Change in Body Composition | 24 weeks
  Assessed via dual x-ray absorptiometry
Change in Quality of Life | 24 weeks
  Assessed via the Short Form-36v2 Health Survey questionnaire
Dietary Adherence | 24 weeks
  Assessed via adherence to prescribed versus measured energy intake assessed by food records
Examine mechanisms related to prebiotic-induced changes in gut microbiota, their metabolic byproducts, and de novo lipogenesis | 24 weeks
  Via investigating gut microbiota shot-gun sequencing and measurement of volatile organic compounds and de novo lipogenesis using deuterium incorporation

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mayengbam S, Raman M, Parnell JA, Eksteen B, Lambert JE, Eller LK, Nicolucci AC, Aktary ML, Reimer RA. Effects of combined prebiotic fiber supplementation and weight loss counseling in adults with metabolic dysfunction-associated steatotic liver disease: a randomized controlled trial. Eur J Nutr. 2025 Apr 2;64(4):144. doi: 10.1007/s00394-025-03660-7. PMID 40172664
- [Derived] Lambert JE, Parnell JA, Eksteen B, Raman M, Bomhof MR, Rioux KP, Madsen KL, Reimer RA. Gut microbiota manipulation with prebiotics in patients with non-alcoholic fatty liver disease: a randomized controlled trial protocol. BMC Gastroenterol. 2015 Dec 3;15:169. doi: 10.1186/s12876-015-0400-5. PMID 26635079